CLINICAL TRIAL: NCT04650607
Title: Phage Safety Cohort Study
Acronym: PHA-SA-CO
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 30032022
Record Dates: First submitted 2020-11-25; First posted 2020-12-02 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2022-05

CONDITIONS: Prosthetic Joint Infection; Severe Infection
Keywords: phage; adverse event; severe infection; compassionate treatment
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — PBMC, serums, plasmas
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PHA SA CO: patients having a severe infection treated by injection of phages, with or without surgery
  Interventions: Other: Adverse event after injection of phages
- PhageRESPONSE: ancillary study : Establish a biobanking of serums, plasmas and PBMC (Peripheral Blood Mononuclear Cells) of patients who have been treated with phage therapy for a bacterial infection.
  Interventions: Other: Adverse event after injection of phages

INTERVENTIONS:
Other: Adverse event after injection of phages — rate and description of adverse event after injection of phages

SUMMARY:
This cohort study aims to describe the adverse events related to the use of bacteriophages to treat serious infections, data from the literature being almost non-existent on this subject.

DETAILED DESCRIPTION:
All potential serious adverse events in compassionate cases will be collected, and classified as potentially related to surgery, to antibiotics, or to phages, with the help of the HCL pharmacovigilance center. In addition, biobanking of pre- and post-treatment blood specimens (bloods, serums and cells) will determine whether phage immunization is implicated in particular adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age or older with a serious infection treated at CRIOAc Lyon by phage therapy
* Patient who did not object to participating in the study
* Patients ayant un poids minimum de 46kg

Exclusion Criteria:

* Patients under guardianship/curatorship
* Patients deprived of liberty
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients having a severe infection treated by injection of phages at the CRIOAC Lyon, Croix-Rousse Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-05-09 (Actual); Primary Completion 2023-10-09 (Estimated); Study Completion 2028-05-09 (Estimated)

PRIMARY OUTCOMES:
type of adverse event | 12 months after the injection of phages
  description of the adverse event
rate of adverse event | 12 months after the injection of phages
  proportion of patient having an avderse event after injection of phages

SECONDARY OUTCOMES:
biobanking PHA SA CO | from before the injection of phages to 6 months after the injection of phages
  to assess the role of immunization induced by phage phages in the occurrence of adverse
biobanking PhageRESPONSE | from before the injection of phages to 6 months after the injection of phages
  Characterize the cellular and humoral immune response in patients with a severe bacterial infection requiring treatment compassionate by bacteriophage

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.crioac-lyon.fr/